CLINICAL TRIAL: NCT02506166
Title: European Sleep Apnea and Sudden CArdiac Death ProjEct
Acronym: ESCAPE-SCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Olomouc (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, doc. MUDr. Miloš Táborský, CSc., FESC, MBA, Chair, Department of Cardiology, University Hospital Olomouc, University Hospital Olomouc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44/15 ESCAPE - SCD
Record Dates: First submitted 2015-07-20; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Sleep Apnea; Sudden Cardiac Death; Heart Failure; Ischemic Cardiomyopathy
Keywords: sleep apnea; sleep disordered breathing; sudden cardiac death; heart failure; ischemic cardiomyopathy; implantable cardioverter-defibrillator (ICD) therapy; cardiac resynchronization therapy (CRT); risk stratification; positive airway pressure therapy; SERVE-HF
MeSH Terms: conditions — Sleep Apnea Syndromes; Death, Sudden, Cardiac; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- No or Mild Sleep Apnea Group (Group 1) (No Intervention): ICM patients with no or mild sleep apnea enrolled in this arm will continue with standard therapy (ICD/CRT-D implant + maximal medical therapy), but will receive no active Positive Airway Pressure (PAP) therapy for sleep apnea treatment. See Part: "Study Population" for more details.
  In all ICM patients enrolled into ESCAPE-SCD Study, the ICD/CRT-D devices will be implanted based on current ESC Guidelines for primary prevention of sudden cardiac death (see Section: "References")
- Obstructive Sleep Apnea - Control Group (Group 2) (No Intervention): ICM patients with predominant obstructive sleep apnea randomised to this arm will receive standard therapy (ICD/CRT-D implant + maximal medical therapy), but no PAP therapy for sleep apnea treatment. See Part: "Study Population" for more details.
- Obstructive Sleep Apnea - Active Group (Group 3) (Active Comparator): ICM patients with predominant obstructive sleep apnea randomised to this arm will receive standard therapy (ICD/CRT-D implant + maximal medical therapy), plus as intervention, all patinets in this group will receive sleep apnea treatment by using PAP device. See Part: "Study Population" for more details.
  Interventions: Device: Positive Airway Pressure Therapy
- Central Sleep Apnea Group (Group 4) (No Intervention): ICM patients with predominant central sleep apnea enrolled in this group will receive standard therapy (ICD/CRT-D implant + maximal medical therapy). Because the SERVE-HF Trial demonstrated a negative effect of predominantly central sleep apnea treatment on cardiovascular mortality in patients with HFrEF by using adaptive servo-ventilation therapy, patients in Group 4 will not receive any PAP therapy for treatment of sleep disordered breathing. See Part: "Study Population" for more details.

INTERVENTIONS:
Device: Positive Airway Pressure Therapy — Positive Airway Pressure Therapy will be used in Group 3 for treatment of predominant obstructive sleep apnea
  Arms: Obstructive Sleep Apnea - Active Group (Group 3)

SUMMARY:
The objective of ESCAPE-SCD Study is assessment of the effect of sleep apnea on sudden cardiac death risk and cardiovascular outcomes in patients with ischemic cardiomyopathy. The ESCAPE - SCD Study will address following specific study questions:

* Is obstructive sleep apnea (OSA) and/or central sleep apnea (CSA) an independent risk factor of sudden cardiac death (SCD) in patients with ischemic cardiomyopathy (ICM) indicated for ICD/CRT-D implant based on current European Society of Cardiology (ESC) Guidelines for primary prevention of sudden cardiac death?
* Can treatment of predominant (>50%) obstructive sleep apnea by appropriate Positive Airway Pressure (PAP) therapy decrease risk of sudden cardiac arrhythmic death in ICM patients?
* Can treatment of predominant (>50%) obstructive sleep apnea by appropriate PAP therapy improve cardiovascular outcomes in ICM patients indicated for ICD/CRT-D implant?
* Does obstructive sleep apnea represent a novel factor that may improve risk stratification of sudden cardiac death and advance identification of those patients that will benefit from ICD/CRT-D therapy?

DETAILED DESCRIPTION:
Detailed Study Description

Purpose:

There is strong evidence that patients with ischemic cardiomyopathy have high cardiovascular mortality, including high risk of sudden cardiac death. Sleep apnea is frequently present in patients after myocardial infarction/with ischemic cardiomyopathy (approximately in 50% of patients).

Both central and obstructive sleep apnea are considered as independent risk factors of worsened prognosis in patients with heart failure with reduced ejection fraction (HFrEF). However, there is no evidence from randomized trials yet providing evidence that sleep apnea is an independent risk factor leading to an increase in cardiovascular mortality, including increased risk of sudden cardiac arrhythmic death in patients with ischemic cardiomyopathy. There are also no data from randomized trials assessing if treatment of sleep apnea by positive airway pressure therapy may improve cardiovascular outcomes in these patients, including reduced risk of sudden cardiac death.

Rationale:

ICD therapy decreases risk of sudden cardiac death in patients with HFrEF, including patients with ICM with left ventricular ejection fraction of <35%. Current ESC Guidelines for implantable cardioverter defibrillator (ICD) therapy for primary prevention of sudden cardiac death in patients with ischemic cardiomyopathy have high sensitivity and high positive predictive value. A limitation of current guidelines is low specificity and low negative predictive value. In real clinical practice, it means that less than 1/3 of patients with heart failure with reduced ejection fraction who get the ICD device for an indication of primary prevention of sudden cardiac death will receive appropriate ICD discharge. The remaining 2/3 of patients have no benefit from ICD implantation, and are exposed to risks of complications resulting from ICD implant, such as inappropriate ICD discharges, lead dislocation, or even life-threatening complications such as infectious endocarditis or myocardial perforation.

Therefore, improvements of stratification criteria allowing better identification of those patients with ICM that will have real benefit from ICD therapy, and improvement of long-term outcomes and cost-benefit of ICD therapy, represent one of the major challenges of modern cardiology.

Previous studies show that sleep apnea increases the risk of sudden cardiac death in the population. In other words, sleep apnea represents a treatable condition which is also a potential risk factor of sudden cardiac death. Some previously non-randomized studies showed that in patients with HFrEF, both obstructive and central sleep apnea may increase risk of sudden cardiac arrhythmic death. Contrary to these observations, recently released preliminary data from the SERVE-HF trial indicate that in patients with HFrEF, treatment of central sleep apnea by adaptive servo-ventilation therapy increases cardiovascular mortality, and responsible mechanisms might include increased risk of sudden cardiac death.

There are several pathophysiological mechanisms by which both obstructive and central sleep apnea may increase risk of sudden cardiac arrhythmic death in ICM patients. Considering the high prevalence of sleep disordered breathing in patients with ICM, sleep apnea represents a modifiable risk factor, where proper treatment may decrease risk of sudden cardiac death and/or improve cardiovascular outcomes in ICM patients. However, randomized studies specifically addressing the role of sleep apnea in risk of sudden cardiac arrhythmic death in ICM patients are needed to clarify the existing controversy and provide information highly needed for routine clinical practice.

Objective

The ESCAPE - SCD Study will address following specific study questions:

* Is obstructive sleep apnea and/or central sleep apnea an independent risk factor of sudden cardiac death (SCD) in patients with ICM indicated for ICD/CRT-D implant based on current ESC Guidelines for primary prevention of sudden cardiac death?
* Can treatment of predominant (>50%) obstructive sleep apnea by appropriate Positive Airway Pressure (PAP) therapy decrease risk of sudden cardiac arrhythmic death in ICM patients?
* Can treatment of predominant (>50%) obstructive sleep apnea by appropriate PAP therapy improve cardiovascular outcomes in ICM patients indicated for ICD/CRT-D implant?
* Does obstructive sleep apnea represent a novel factor that may improve risk stratification of sudden cardiac death and advance identification of those patients that will benefit from ICD/CRT-D therapy?

Study Design:

Prospective, randomized, international multi-centric study.

Study Population:

900 patients with ICM indicated for ICD/CRT-D implant based on 2012 and 2013 ESC Guidelines for primary prevention of sudden cardiac death (see Section: "References") will be enrolled in this study. A sleep study will be performed in each of the subjects and based on results patients will be divided to 4 Groups.

• No or Mild Sleep Apnea Group (Group 1): Patients with no or mild sleep apnea will continue with standard therapy (ICD/CRT-D implant + maximal medical therapy).

Patients with moderate and severe predominant obstructive sleep apnea (AHI >15) will be randomized in 1:1 ratio to

* Obstructive Sleep Apnea - Control Group (Group 2) - patients with predominant obstructive sleep apnea that will receive standard therapy (ICD/CRT-D implant + maximal medical therapy), but no PAP therapy for sleep apnea treatment and to
* Obstructive Sleep Apnea - Active Group (Group 3) - patients with predominant obstructive sleep apnea that will receive standard therapy (ICD/CRT-D implant + maximal medical therapy), plus, as intervention, sleep apnea treatment by using PAP therapy.
* Central Sleep Apnea Group (Group 4) - patients with predominant central sleep apnea that will receive standard therapy (ICD/CRT-D implant + maximal medical therapy). Because the SERVE-HF Trial demonstrated a negative effect of predominantly central sleep apnea treatment on cardiovascular mortality in patients with HFrEF by using adaptive servo-ventilation therapy, patients in Group 4 will not receive any PAP therapy for treatment of sleep disordered breathing and will be followed.

Distribution of Patient Population among Study Group:

Based on data derived from our pilot study, approximately 60% of patients with ischemic cardiomyopathy indicated for ICD/CRT-D implant for primary prevention of sudden cardiac death have undiagnosed moderate or severe sleep apnea. Therefore, we expect the following distribution of patients among patients' groups: Group 1: n=400 patients; Group 2: n=200 patients; Group 3: n=200, Group 4: n=100 patients.

Primary and secondary goals:

Primary goal:

* Assessment of sleep apnea and its treatment on risk of sudden cardiac arrhythmic death by assessing the number of appropriate ICD/CRT-D discharges for each of the groups

Secondary goals:

* Assessment of the effect of sleep apnea and OSA treatment on cardiovascular mortality and morbidity by assessing MACE (Major Adverse Cardiovascular Events)
* Assessment of incidence of complications resulting from ICD/CRT-D therapy among study groups
* Assessment of sleep apnea as a novel factor that may improve risk stratification of sudden cardiac death and advance identification of those patients that will benefit from ICD/CRT-D therapy.
* Assessment of sleep apnea treatment on systolic and diastolic functions and neurohumoral profile
* Assessment of prevalence of sleep apnea and its severity among study population

Eligibility

Ages Eligible for Study: 18 Years and older Genders Eligible for Study: Both Accepts Healthy Volunteers: No

Technologies used for sleep apnea treatment It is planned to use the Airsense 10 Autoset (AutoCPAP) and Aircurve 10 CS Pacewave (AutoASV) RESMED devices for sleep disordered breathing treatment in Group 3 with sleep apnea treatment telemonitoring option.

Technologies used for detection of life-threatening ventricular arrhythmias:

Most advanced ICD/CRT-D technologies allowing telemonitoring detection of cardiac arrhythmias will be used in as many patients as possible who are enrolled into this study.

Study Timeline:

* Study initiation: January 2016
* Patient enrollment: March 2016 - December 2017
* Average follow-up: 36 months
* End of follow-up: December 2019
* Data analysis: January-December 2021
* Estimated publication of final results: 2022

Study Co-Principal Investigators (listed alphabetically): Assoc. Prof. Tomas Kara, MD, PhD, Prof. Virend K. Somers, MD, DPhil., Prof. Milos Taborsky, MD, PhD

Study sponsors:

Investigator Initiated Trial.

Contacts and locations:

Coordinating center:

Department of Cardiovascular Diseases University Hospital Olomouc I.P. Pavlova 6 779 00 Olomouc, Czech Republic Phone.: +420 58 588 3201 Fax: +420 58 588 2500

Summary:

This would be the very first randomized study assessing the effect of predominantly obstructive sleep apnea treatment on risk of sudden cardiac death and cardiovascular outcomes in patients with ischemic cardiomyopathy. The study will also address important questions related to improvement of selection of patients that may benefit from ICD/CRT-D therapy. We have solid evidence from our pilot data that addition of sleep disordered breathing screening and treatment may improve the selection of patients with ischemic cardiomyopathy that can benefit from ICD therapy, including improvement their long-term outcomes. Use of technologies for telemonitoring of efficiency of sleep disordered breathing treatment and occurrence of cardiac arrhythmias will increase the scientific strength of the study and will explore the benefit of use of telemonitoring technologies in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Patients with ICM indicated for ICD/CRT-D implant based on current ESC Guidelines for primary prevention of sudden cardiac death

Exclusion Criteria:

* Previously diagnosed sleep apnea CPAP, BiPAP or ASV treatment
* Patients with previously implanted ICD/CRT-D device indicated for device replacement
* Uncontrolled hypertension
* Severe valvular heart disease/dysfunction with exception of ischemic and functional mitral regurgitation
* Acute coronary syndrome or acute cardiac decompensation in 4 weeks before ICD/CRT-D implant
* Expected indication of heart transplant in period of 12 months or less after ICD/CRT-D implant
* Expected cardiac surgery or percutaneous coronary intervention in period of 12 months or less after ICD/CRT-D implant
* Severe pulmonary diseases
* Rejection of participation in the study
* Pregnancy
* Age of 80 years and higher in time of ICD/CRT-D implant

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of sleep apnea and its treatment on risk of sudden cardiac arrhythmic death by assessing the number of appropriate ICD/CRT-D discharges for each of the groups | 36 months

SECONDARY OUTCOMES:
Assessment of the effect of sleep apnea and OSA treatment on cardiovascular mortality and morbidity by assessing the incidence of MACE (Major Adverse Cardiovascular Events) | 36 months
  MACE will be particularly assessed as: death of any cardiovascular origin, heart transplantation, myocardial revascularization, non-fatal stroke, hospitalization for heart failure progression, hospitalization for any cardiovascular origin
Assessment of incidence of complications resulting from ICD/CRT-D therapy among study groups | 36 months
  Incidence of inappropriate ICD discharges, lead dislocation, device malfunction, infectious endocarditis, myocardial perforation will be particularly compared among groups.
Assessment of sleep apnea as a novel factor that may improve risk stratification of sudden cardiac death and advance identification of those patients that will benefit from ICD/CRT-D therapy | 36 months
  Correlation between apnea hypopnea index and incidence of appropriate ICD/CRT-D discharges will be compared among groups
Assessment of effect of sleep apnea treatment on systolic and diastolic functions and neurohumoral profile | 36 months
  Ejection fraction will be used to determine systolic function. Standard criteria for diastolic dysfunction measurement will be used
Assessment of prevalence of sleep apnea among study population | Time of enrollenment
  Apnea-hypopnea index will be used to determine the severity of sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Kara, Assoc. Prof., MD, PhD, Principal Investigator — University Hospital Olomouc; Virend K Somers, Prof., MD, DPhil, Principal Investigator — Mayo Clinic; Milos Taborsky, Prof., MD, PhD, FESC, Principal Investigator — University Hospital Olomouc

REFERENCES:
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE; ESC Committee for Practice Guidelines (CPG); Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Kirchhof P, Blomstrom-Lundqvist C, Badano LP, Aliyev F, Bansch D, Baumgartner H, Bsata W, Buser P, Charron P, Daubert JC, Dobreanu D, Faerestrand S, Hasdai D, Hoes AW, Le Heuzey JY, Mavrakis H, McDonagh T, Merino JL, Nawar MM, Nielsen JC, Pieske B, Poposka L, Ruschitzka F, Tendera M, Van Gelder IC, Wilson CM. 2013 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: the Task Force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Eur Heart J. 2013 Aug;34(29):2281-329. doi: 10.1093/eurheartj/eht150. Epub 2013 Jun 24. No abstract available. PMID 23801822